CLINICAL TRIAL: NCT03781661
Title: Providing Patients With Extended Information and Examination Results Immediately After a Diagnostic CT of the Coronary Arteries
Brief Title: Providing Patient Information and CT Examination Results
Acronym: INFOCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/1380
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2018-08

CONDITIONS: Chest Pain; Nonmalignant Condition
Keywords: Non coronary Chest Pain; Extended Information; Normal Examination Result; Coronar Computed Tomography Angiography; CCTA; Calcium score; Diagnostic Examination; Patient Satisfaction; Normal Coronary Arteries
MeSH Terms: conditions — Chest Pain; Precancerous Conditions; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Experimental randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The participants in the intervention group will be provided with extended information of the advantages of the CT examination of the heart's arteries. This will be given to the participants both orally and written in form of a leaflet. In addition will they be given the opportunity for a visual go-through of their own calcium score images. After this they will be informed of the normal examination result.
  Interventions: Other: Extended information
- Control group (No Intervention): Control Group receives standard care.

INTERVENTIONS:
Other: Extended information — The extended information consists out of an information leaflet and a visual go-through of the participants calcium score images. The patients are then given the normal examination result.
  Arms: Intervention Group

SUMMARY:
Chest pain is a common cause of visits in the Emergency Room and General Practice, and is most commonly connected as a symptom of coronary disease, as for instance angina pectoris and acute myocardial infarct. Approximately 75-80% of these patients are not diagnosed with coronary disease or other cardiac findings. However, many of these patients still report chest pain and worries about cardiac disease.

This study is based on patients that are referred to a CT-examination of the coronary arteries on the background of chest pain, where the CT-examination shows normal coronary arteries.

The study aims to evaluate whether providing an intervention to this group of patients has an effect on patient satisfaction, patient's worry of cardiac disease and incidence of chest pain.

The intervention group will be compared with a similar group going through the same CT-examination, but is receiving the examination result from their regular general practitioner (RGP), which is considered standard care.

The hypothesis is that patients with chest pain with no coronary findings receiving extended information before getting the normal examination results experience a better patient satisfaction than those receiving the examination result from their RGP.

DETAILED DESCRIPTION:
This study is a randomized controlled study. Eligible patients going through a CT-examination of the heart's coronary arteries, Coronary CT Angiogram (CCTA) will after an informed consent be randomized into two groups, either the intervention group or standard care.

The intervention consists of extended information regarding the benefits of doing a CCTA, thereby emphasising the specificity and accuracy of the CCTA's ability to exclude coronary disease. After this, there will be given an opportunity of a visual go-through and explanation of CT-images. Then they will be informed of the examination result that shows normal coronary arteries.

Follow up is planned after one month, six months and twelve months, where the participants receive the same questionnaire as at baseline to fill out and return. The questionnaire consists of Seattle Angina Questionnaire and RAND-12, in addition to social demographic and clinical data, such as sex, height, weight and current medication.

ELIGIBILITY:
Inclusion Criteria:

* ability to speak and read Norwegian fluently
* competent to give informed consent
* referred from cardiologist
* experienced chest pain
* Calcium score = 0 and CCTA must show normal coronary arteries
* received information letter on ongoing research in the Heart department of Haukeland University Hospital

Exclusion Criteria:

* admitted patients
* heart disease or coronary anomalies shown on the CCTA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction: Seattle Angina Questionnaire | 1 month
  Our primary outcome is to examine whether patients with chest pain with normal coronary arteries experience greater satisfaction with their treatment if they receive extended information and the examination results immediately after the CT examination than those who receive the examination result from their RGP.
  This is measured with 2 single items in Seattle Angina Questionnaire regarding satisfaction with treatment. Values range from 1-5, 1 is the lowest level of satisfaction, and 5 is the highest level of satisfaction. Greater satisfaction with treatment will be defined by a higher score at follow-up after 1 month.
  In addition, there is a separate question of patients' trust in the CT examination measured with a VAS-scale , ranging from 1-10, 1 represents lowest possible degree of trust, and 10 represents highest possible degree of trust. Greater trust in the CT-examination is defined by higher scores at follow-up after 1 month.

SECONDARY OUTCOMES:
Worry of having heart disease | 1 month, 6 months, 12 months
  To examine if patients report less worry of having a heart attack or sudden death after having a CT examination of the heart's arteries, when receiving extended information and the normal examination result immediately after the CT examination.
  This is measured with a single item in Seattle Angina Questionnaire regarding worry of having heart attack or die suddenly. Values range from 1-5, 1 represents "worry all the time" and 5 represents "never worry". Less worry of having a heart attack or die suddenly will be defined by higher scores at follow-up after 1, 6 and 12 months.
Incidence of chest pain | 1 month, 6 months, 12 months
  To examine if patients with chest pain with normal coronary arteries report less chest pain and/or less use of health care services if they receive extended information and the examination results immediately after the CT examination compared to those who receive the examination result from their RGP.
  This is measured with 2 single items in Seattle Angina Questionnaire. One item regards limitations in everyday activities because of chest pain. Values range from 1-5, 1 represents lowest level, and 5 represents highest level of function. The second item is about incidence of chest pain the last week. Values range from 1-5, 1 represents high incidence of chest pain and 5 represents no chest pain. Less chest pain is associated with higher scores at all times of follow up, compared to baseline.
  In addition, clinical data regarding participants use of primary and secondary health care the last 4 weeks is collected at all times of follow-up and is compared to baseline data.
Patient satisfaction: Seattle Angina Questionnaire | 6 months, 12 months
  To examine whether patients with chest pain with normal coronary arteries experience greater satisfaction with their treatment if they receive extended information and the examination results immediately after the CT examination than those who receive the examination result from their RGP.
  This is measured with 2 single items in Seattle Angina Questionnaire regarding satisfaction with treatment. Values range from 1-5, 1 is the lowest level of satisfaction, and 5 is the highest level of satisfaction. Greater satisfaction with treatment will be defined by a higher score at follow-up after 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tone M Norekvaal, Professor, Principal Investigator — University of Bergen
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krohn IL, Rygh CB, Larsen TH, Wentzel-Larsen T, Norekval TM. Effect of radiographer-led intervention on reassurance, treatment satisfaction, and recurring chest pain in patients with a normal coronary computed tomography angiography-a randomized controlled trial. Eur J Cardiovasc Nurs. 2022 Jun 2;21(4):318-324. doi: 10.1093/eurjcn/zvab064. PMID 34601588